CLINICAL TRIAL: NCT03563235
Title: Clinical Study on Treatment of Postmenopausal Osteoporosis (Kidney Deficiency and Blood Stasis Syndrome) With Xulin Jiangu Granules
Acronym: CSOPOPWXJG
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Academy of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018R1035-4
Record Dates: First submitted 2018-05-31; First posted 2018-06-20 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Postmenopausal Osteoporoses
Keywords: Osteoporosis; kidney deficiency and blood stasis syndrome; Xuling Jiangu Granules
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis | interventions — Calcitriol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xulin Jiangu granules (Experimental): Xulin Jiangu granule 15g tablet by mouth every 6 hour for 6 months
  Interventions: Drug: Xulin Jiangu granules; Drug: Calcitriol capsules
- Calcitriol capsules (Active Comparator): Calcitriol capsules tablets 0.25 ug by mouth every 6 hour for 6 months
  Interventions: Drug: Xulin Jiangu granules; Drug: Calcitriol capsules

INTERVENTIONS:
Drug: Xulin Jiangu granules — Xulin Jiangu granules tablets
Drug: Calcitriol capsules — Calcitriol capsules tablets

SUMMARY:
Osteoporosis is a common senile disease with a high incidence. The Chinese medicine differentiation treatment has small side effects and can be taken for a long time, which has certain advantages. This project adopts the experience of the person in charge of the project-Xulin Jiangu Granules and clinically collects patients with postmenopausal osteoporosis (kidney deficiency and blood stasis syndrome).

DETAILED DESCRIPTION:
Randomized control method was used to observe the clinical efficacy of the treatment of postmenopausal osteoporosis (kidney deficiency and blood stasis syndrome) with jiujian jiangu granules, combined with the gene expression of bone metabolism markers BALP, PINP, TRACP and S-CTX, and RANK, RANKL and OPG Detection, compared with the control group of ossification trihydrate capsules, to explore the mechanism of the treatment of postmenopausal osteoporosis by the continued Xulin Jiangu granules, and lay the foundation for the development of new drugs.

ELIGIBILITY:
Inclusion Criteria:

* at least 2 years prior and met the diagnostic criteria for osteoporosis according to the "clinical practice guidelines of traditional medicine for primary osteoporosis
* met the CM diagnostic criteria according to "Syndrome Differentiation in Modern Research of Traditional Chinese Medicine

Exclusion Criteria:

* patients who did not meet the diagnostic criteria for osteoporosis or CM standards
* patients with rheumatoid arthritis, diabetes, secondary osteoporosis due to hyperthyroidism, and severe cardiovascular or cerebrovascular diseases
* patients with abnormal liver and/or Shen function test results
* patients with osteoporosis who had received treatment with CM within the last month, hormone replacement therapy and calcitonin within the past three months, or bisphosphonates for 15 consecutive days within the past 6 months.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Bone density（BMD） | Xulin Jiangu treats for up to six months
  BMD is the gold standard of oeteoporosis

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Academy of Trational Chiness Medicine, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No